CLINICAL TRIAL: NCT05997485
Title: A Retrospective Observational Non-Interventional Study (NIS) to Assess Patient Characteristics Among COVID-19 Patients Receiving Treatment With Nirmatrelvir/Ritonavir (PAXLOVIDTM) in Morocco.
Brief Title: A Study to Learn About the Patients With COVID-19 Prescribed Paxlovid in Morocco
Status: Withdrawn | Type: Observational
Why Stopped: The study was prematurely discontinued due to the substantial delay in initiation the study. This decision was not due to major safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671060
Record Dates: First submitted 2023-08-15; First posted 2023-08-18 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Drug Treatment
Keywords: Treatment; Covid Patient; Paxlovid; Morocco
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Participants receiving Paxlovid Treatment: Patients administered oral Paxlovid as prescribed according to national Morocco treatment guidelines for Covid.
  Interventions: Drug: Nirmatrelvir/Ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/Ritonavir — Patients administered oral Paxlovid as prescribed according to national Morocco treatment guidelines for Covid.
  Other Names: Paxlovid

SUMMARY:
The purpose of this study is to collect information on the:

* general information of a group of people such as their age, sex, and other facts.
* clinical information of the patients such as any other illness before having COVID 19.

In adult patients with COVID-19 who have been prescribed nirmatrelvir and ritonavir treatment.

This study will be conducted in Morocco. The study will capture information of the adult COVID-19 outpatients and inpatients who have been prescribed nirmatrelvir, ritonavir treatment. The inpatients will be admitted in the hospital for other reasons than COVID-19.

This study will have about 150 patients. The study will involve collection of patient information from medical records. The information collected can be either from papers or from computers.

The study will include patient information of those who:

* are confirmed to have COVID-19 infection during the study period from 01 June 2022 to 30 June 2023.
* are 18 years of age or older.
* are prescribed Nirmatrelvir and ritonavir. This study will help to inform decision-making on use of Paxlovid at the national level.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection during the study period from 01 June 2022 to 30 June 2023
* Nirmatrelvir, ritonavir written prescription

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants treated with Paxlovid in single center in Morocco.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographical Characteristics of Participants | Approximately 01 June 2022 through 30 June 2023
Clinical Characteristics of Participants | Approximately 01 June 2022 through 30 June 2023
Number of Participants with Pre-existing Comorbidities | Approximately 01 June 2022 through 30 June 2023

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.